CLINICAL TRIAL: NCT03575299
Title: Clinical Study on Adoptive Treatment of Multidrug Resistant Pulmonary Tuberculosis With Allogeneic γδT Cells
Brief Title: Clinical Study on Adoptive Treatment of MDR-TB With Allogeneic γδT Cells
Acronym: MDR-TB
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Zhinan Yin, Ph.D. (Other)
Collaborators: Shenzhen Third People's Hospital (Other)
Responsible Party: Sponsor-Investigator, Zhinan Yin, Ph.D., Dean of Biomedical Translational Research Institute，jinan University, Jinan University Guangzhou
Organization: Jinan University Guangzhou (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: GDT-MDR-TB-069
Record Dates: First submitted 2018-06-19; First posted 2018-07-02 (Actual); Last update posted 2018-07-02 (Actual); Status verified 2018-06

CONDITIONS: Multi-drug Resistant Tuberculosis
Keywords: MDR-TB; Allogeneic γδT cells; adoptive treatment
MeSH Terms: conditions — Tuberculosis, Multidrug-Resistant

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Study group (Experimental): Patients will be treated with anti-tuberculosis drugs, and meanwhile will be treated with Allogeneic γδT cells.
  Interventions: Biological: The adoptive treatment of allogeneic γδT cells; Drug: Conventional treatment
- Control Group (Placebo Comparator): Patients will be treated with anti-tuberculosis drugs, and meanwhile will not be treated with allogeneic γδT cells.
  Interventions: Other: Control; Drug: Conventional treatment

INTERVENTIONS:
Biological: The adoptive treatment of allogeneic γδT cells — Allogeneic γδT cells will be administered to patients with MDR-TB every two weeks, for 12 times in a total of 6 months.
  Arms: Study group
Other: Control — No allogeneic γδT cells will be administered to patients with MDR-TB.
  Arms: Control Group
Drug: Conventional treatment — Patients will be treated with anti-tuberculosis drugs throughout the entire process of the study.

SUMMARY:
Brief summary: Allogeneic γδT cells from healthy donor will be administrated intravenously to patients with the MDR-TB，and then the safety and efficacy of γδT cells will be evaluated.

DETAILED DESCRIPTION:
All patients with multi-drug resistant pulmonary tuberculosis will be assigned into 2 groups(study group and control group)，both groups will receive conventional treatment. Allogeneic γδT cell will be administrated intravenously to patients in the study group (but not the control group) every two weeks for 6 months

ELIGIBILITY:
Inclusion Criteria:

1. Aged 18-50 years old, male or female;
2. Informed consent;
3. Patients with multidrug-resistant tuberculosis diagnosed by positive sputum smear and tubercle bacillus culture.

Exclusion Criteria:

1. AIDS, hepatitis B and other viruses, bacterial infections;
2. Patients with other diseases such as diabetes, cancer, hypertension, coronary heart disease, endocrine system diseases, mental diseases, neurological diseases, and vascular circulatory diseases;
3. Others After being evaluated by clinicians participating in this project, it is not suitable to participate in immune cell therapy;
4. Those who do not agree to be included.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 45 (Estimated)
Dates: Start 2018-06-01 (Actual); Primary Completion 2021-06-30 (Estimated); Study Completion 2021-12-31 (Estimated)

PRIMARY OUTCOMES:
sputum smear | 6 months
  The sputum specimens will be collected biweekly in the first 2 months and bimonthly thereafter for sputum smear to study the time (months) of the sputum conversion. The sputum conversation rate will be analyzed at the end of study.

SECONDARY OUTCOMES:
Sputum tubercle bacillus culture | 6 months
  The sputum specimens will be collected for culture to detect the TB biweekly in the first 2 months and bimonthly thereafter to study the time (months) of the sputum conversion. The sputum conversation rate will be analyzed at the end of study.
Fecal microbiome analysis | 6 months
  The faeces will be taken to study fecal microbiome changes biweekly in the first 2 months, and monthly thereafter.
Assessment of immune function | 6 months
  Peripheral blood will be collected for assessment of immune system function every time before the administration of allogeneic γδT cells .

CONTACTS AND LOCATIONS:
Overall Officials: Guofang Deng, Master, Principal Investigator — Partner
Locations (1):
- Shenzhen Third People's Hospital, Shenzhen, Guangdong, China

REFERENCES:
- [Derived] Liang J, Fu L, Li M, Chen Y, Wang Y, Lin Y, Zhang H, Xu Y, Qin L, Liu J, Wang W, Hao J, Liu S, Zhang P, Lin L, Alnaggar M, Zhou J, Zhou L, Guo H, Wang Z, Liu L, Deng G, Zhang G, Wu Y, Yin Z. Allogeneic Vgamma9Vdelta2 T-Cell Therapy Promotes Pulmonary Lesion Repair: An Open-Label, Single-Arm Pilot Study in Patients With Multidrug-Resistant Tuberculosis. Front Immunol. 2021 Dec 15;12:756495. doi: 10.3389/fimmu.2021.756495. eCollection 2021. PMID 34975844